CLINICAL TRIAL: NCT02560259
Title: The Role of Referred Pain From the Retro Trochanteric Region in Patients With Knee Pain. Prevalence, Interpretation and Management: A Randomized Controlled Study
Brief Title: The Role of Referred Pain From the Retro Trochanteric Region in Patients With Knee Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital of North Norway (Other)
Responsible Party: Principal Investigator, Oddmund Johansen, Professor, University Hospital of North Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/157(REK)
Record Dates: First submitted 2015-05-11; First posted 2015-09-25 (Estimated); Last update posted 2015-09-25 (Estimated); Status verified 2015-09

CONDITIONS: Referred Pain
Keywords: knee pain
MeSH Terms: conditions — Pain, Referred | interventions — Physical Therapy Modalities; Conservative Treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Physiotherapy Group (Active Comparator): Physiotherapy
  Interventions: Other: Physiotherapy
- Conservative group (Placebo Comparator): Conservative treatment
  Interventions: Other: Conservative treatment

INTERVENTIONS:
Other: Physiotherapy — Physiotherapy
  Arms: Physiotherapy Group
Other: Conservative treatment — Conservative treatment
  Arms: Conservative group

SUMMARY:
The role of referred pain from the retro trochanteric region, in patients with knee pain. Defining and quantifying this sub group of knee patients in the investigators list of refered knee patients. Evaluating the effect of treatment. A randomized trial.

DETAILED DESCRIPTION:
Knee pain is a great problem in the society. Besides obvious and known causes, for which there are increasing understanding and ways to treat, there is still a rather large group of patients in which the symptoms are not easily understood and harder to treat.

This group is often characterized by having symptoms ranging from months to years, having seen several physicians, gone through several x-rays/mri´s, and various treatment with no help.

The investigators find ever more suspicion towards specific mechanisms in the hip region as a source of knee pain. It is well known in pediatric medicine that children with serious disease in the hip often debut with knee pain. This relationship is not so well established in adults.

Pain in the lower extremity can arise from inflammation or strain of the retro trochanteric muscles, and/or more indirectly if these processes impact the sciatic nerve. The later explanation is commonly known as the piriformis syndrome.

Professor Oddmund Johansen has studied this type of pain extensively. In the later years he has found interest in patients with knee pain.

These patients will often have pain with deep palpation to the posterior hip region, when tightening the hip rotators with flexion and adduction, and they will often respond with pain relief, within minutes, when local anesthesia is placed on the distal attachment of the hip rotators on the posterior margin of the greater trochanter. Afterwards, lasting pain relief can be seen with a specified stretching regiment for these muscles.

The investigators will recruit suiting patients from a knee referral list. Inclusion will be based on clinical examination and whether they respond to the injection. After inclusion they will be scored with pain and quality of life forms, randomised in two groups, one with a stretching regime and one with conservative and symptomatic treatment.

There is interest in defining and quantifying this sub group of knee patients. They will be followed up after 3 months, with a new examination and scoring to evaluate the effect of the intervention.

The study will examine how the patients react and comply with the proposed diagnosis and treatment. A cost analysis will also be considered.

ELIGIBILITY:
Inclusion Criteria:

* Knee pain
* Failure to understand the pain with more conventional diagnosis
* Symptoms and retrotrochanteric pain with examination
* Pain relief with retro trochanteric local anaesthetic injection

Exclusion Criteria:

* Mental illness
* Failure to cooperate
* Not adequate Norwegian language skills
* Other well known disease explaining symptoms

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Pain on VAS score | At 3 months
  0 no pain, 10 worst possible pain

SECONDARY OUTCOMES:
KOOS score subscales Pain | At 3 months
  Standard scoring on the KOOS subscale of pain
KOOS score subscale Symptoms | At 3 months
  Standard scoring on the KOOS subscale of symptoms
KOOS score subscale Function in daily living | At 3 months
  Standard scoring on the KOOS subscale of Function of daily living
KOOS score subscale Knee-Related Quality of Life | At 3 months
  Standard scoring on the KOOS subscale of Knee-Related Quality of Life
KOOS score subscale Function in Sports and Recreation | At 3 months
  Standard scoring on the KOOS subscale of Function in Sports and Recreation

OTHER OUTCOMES:
Working full time the last week | At 3months
  Response yes or no to question if the participant worked full time last week

CONTACTS AND LOCATIONS:
Overall Officials: Oddmund Johansen, Professor, Principal Investigator — University Hospital og North Nprway, ortopedic department
Locations (1):
- University Hospital of Northern Norway, Tromsø, Norway

REFERENCES:
- [Result] Meknas K, Kartus J, Letto JI, Flaten M, Johansen O. A 5-year prospective study of non-surgical treatment of retro-trochanteric pain. Knee Surg Sports Traumatol Arthrosc. 2009 Aug;17(8):996-1002. doi: 10.1007/s00167-009-0750-z. Epub 2009 Mar 5. PMID 19263036
- [Result] Meknas K, Johansen O, Kartus J. Retro-trochanteric sciatica-like pain: current concept. Knee Surg Sports Traumatol Arthrosc. 2011 Nov;19(11):1971-85. doi: 10.1007/s00167-011-1573-2. Epub 2011 Jun 16. PMID 21678093
- [Result] Meknas K, Kartus J, Letto JI, Christensen A, Johansen O. Surgical release of the internal obturator tendon for the treatment of retro-trochanteric pain syndrome: a prospective randomized study, with long-term follow-up. Knee Surg Sports Traumatol Arthrosc. 2009 Oct;17(10):1249-56. doi: 10.1007/s00167-009-0787-z. Epub 2009 Apr 18. PMID 19396428
- [Result] Meknas K, Christensen A, Johansen O. The internal obturator muscle may cause sciatic pain. Pain. 2003 Jul;104(1-2):375-80. doi: 10.1016/s0304-3959(03)00045-9. PMID 12855348